CLINICAL TRIAL: NCT03882281
Title: A Randomized, Open, Double-crossing Trial to Evaluate the Effect of Fasting or High-fat Meals on the Pharmacokinetics of Single Oral Administration of HQP1351 Tablets on an Empty Stomach or a High-fat Meal in Patients With Chronic Myeloid Leukemia
Brief Title: Pharmacokinetics Profiles of HQP1351 Under Fasting and High-fat Meals in Patients With Chronic Myeloid Leukemia
Acronym: CML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: HealthQuest Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351LC104
Record Dates: First submitted 2019-03-12; First posted 2019-03-20 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
Keywords: Chronic Myeloid Leukemia, Chronic Phase; HQP1351
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): Subjects in the group A will be given HQP1351 after fasting meal on Day 1. Then after a seven-day of cleaning time, subjects in the group A will be given HQP1351 after 30 minutes of high-fat meal on Day 8.
  Interventions: Drug: HQP1351
- B group (Experimental): Subjects in the group B will be given HQP1351 after 30 minutes of high-fat meal on Day 1. Then after a seven-day of cleaning time, subjects in the group B will be given HQP1351 after fasting meal on Day 8.
  Interventions: Drug: HQP1351

INTERVENTIONS:
Drug: HQP1351 — Orally, single dose of 30mg on day 1 and day 8.

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of HQP1351 in participants with resistant chronic myeloid leukemia (CML) in chronic phase (CP) after high-fat and fasting meals separately（Selection of high-fat meal spectrum：《The Food - Effect Bioavailability and Fed Bioequivalence Studies》high fat diet should be 800-1000 kcal heat.).

DETAILED DESCRIPTION:
The drug being test in this study is HQP1351，the study will characterize the pharmacokinetics of HQP1351 in participants with resistant chronic myeloid leukemia（CML）in chronic phase（CP）after high-fat meal and fasting meal separately at a dose of 30mg，single-dose. The study will enroll 12 subjects totally and be randomly divided into 2 groups（A group and B group）. Every group will have 6 subjects. The experiment is divided into two periods，in period 1, subjects in the group A will be given HQP1351 30mg after fasting meal，and the group B will be given HQP1351 30mg after 30 minutes of high-fat meal. Then after a seven-day of cleaning time the two groups of subjects took the drug interchangeably in the period 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients age 18-55 years old.
2. CML Patients in CP with Ph-positive or BCR/ABL-positive.
3. Previously treated with and or developed resistance / intolerance to second generation tyrosine kinase inhibitors (TKIs) (dasatinib，nilotinib）or，been identified to have the T315I mutation at any time during treatment.
4. Ability to understand and willingness to sign a written informed consent form. The consent form must be signed by the patient prior to any study-specific procedures.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
6. Predicted life expectancy of ≥3 months.
7. Organ function as indicated by the following laboratory indicators must be met:

   * Hemoglobin ≥8.0g/dL.
   * White blood cell count ≥ 3.0×10^9/L, neutrophil count≥ 1.5 x 10^9/L.
   * Platelet count ≥ 75×10^9/L.
   * Serum creatinine ≤ 1.5×upper limit of normal (ULN) or 24 hours calculated creatinine clearance ≥ 50ml/min when serum creatinine >1.5×ULN.
   * Serum albumin≥ 3.0 g/dL.
   * Total bilirubin ≤ 1.5 x ULN.
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN of institution's normal range.
   * Lipase≤1.5×ULN, Amylase≤1.5×ULN.
   * Prothrombin time (PT), activated partial thromboplastin time (APTT), INR≤1.5×ULN.
8. Cardiac function index: ejection fraction (EF) > 50%.
9. Corrected QT interval (QTc) interval on electrocardiogram (ECG) evaluation: QTc≤450ms in males or ≤470ms in females.
10. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential and their partners throughout the treatment period and for at least 120 days following the last dose of study drug.
11. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Received cytotoxic chemotherapy or radiotherapy within 28 days, interferon or cytarabine within 14 days, any investigational therapy within 14 days prior to the first dose of study drug, or have not recovered (> grade 1 by NCI CTCAE v 4.03) from adverse events (AEs ) (except alopecia) due to agents previously administered.
2. Require concurrent treatment with drugs that may have interactions with the study drug.
3. Have previously been treated with ponatinib (or drugs of similar composition).
4. Absorption disorder syndrome or other diseases affecting oral drug absorption.
5. Have any history of heart or vascular disease, such as hypertension (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90mmHg), or take medications that are known to cause prolonged ECG QT interval.
6. Mean pulmonary artery pressure >25 mmHg.
7. Have a history of serious cardiovascular diseases during the previous treatment of chronic myeloid leukemia with TKI.
8. Underwent autologous or allogeneic stem cell transplant.
9. Abnormal coagulation function，or have a bleeding disorder within 3 months before first administration.
10. Underwent major surgery (with the exception of minor surgical procedures, such as placement or bone marrow biopsy) with 14 days prior to first dose of study drug.
11. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy.
12. Have active nervous system (CNS) disease as evidence by cytology or pathology. In the absence of clinical CNS disease, lumbar puncture is not required.
13. History of primary malignancy (cured for more than 5 years, completely resected superficial skin cancer other than melanoma, adequately treated in-situ cancer, or controlled prostate cancer will not be considered exclusionary).
14. Active symptomatic infection.
15. Known to be allergic to study drug ingredients or their analogues.
16. Are pregnant or lactating or expecting pregnancy during the study program.
17. Suffer from any condition or illness that, in the opinion of the Investigator or the sponsor, would compromise patient safety or interfere with the evaluation of the safety of the study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2019-11-16 (Actual)

PRIMARY OUTCOMES:
Area under the curve from the time of dosing to infinity [AUC(0-inf)] | 1-5 days after every drug administration
  Area under the plasma concentration-time curve from time zero extrapolated to infinity time of HQP1351.
Area under the curve from the time of dosing to the last measurable concentration [AUC(0-last)] | 1-5 days after every drug administration
  Area under the plasma concentration-time curve from time zero to the last measurable time point of HQP1351.
Percentage of AUC(0-inf)_obs due to extrapolation from the last measurable time point to infinity (AUC_%Extrap) | 1-5 days after every drug administration
  Percentage of area under the concentration time curve from time zero extrapolated to infinite time obtained by extrapolation of HQP1351.
Maximum observed concentration (Cmax) | 1-5 days after every drug administration
  Maximum observed plasma concentration of HQP1351.
Time of maximum observed concentration (Tmax) | 1-5 days after every drug administration
  Time to maximum observed plasma concentration of HQP1351.
Terminal elimination half life (T1/2) | 1-5 days after every drug administration
  Terminal elimination half life (T1/2) is defined as the duration until observation of half of the maximum concentration of HQP1351.
Total body clearance for extravascular administration (CL/F) | 1-5 days after every drug administration
  Apparent clearance of HQP1351 following oral dosing. Clearance of a drug is a measure of rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose of HQP1351 (apparent oral clearance) is influenced by the fraction of dose absorbed.
Volume of distribution based on the terminal phase for extravascular administration (Vz/F) | 1-5 days after every drug administration
  Apparent volume of distribution of HQP1351. Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution of HQP1351 after oral dose (Vz/F) is influenced by the fraction absorbed.

SECONDARY OUTCOMES:
Incidence of toxicity | up to 12 days
  Incidence of toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: QIAN JIANG, Professor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China